CLINICAL TRIAL: NCT03906227
Title: Tailoring Maintenance Therapy to CD5+ Regulatory B Cell Recovery in ANCA Vasculitis
Brief Title: Tailoring Maintenance Therapy to Cluster of Differentiation 5 Positive (CD5+) Regulatory B Cell Recovery in ANCA Vasculitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study recruitment terminated due to lack of funding.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-2015; 5P01DK058335-18 (NIH)
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-05

CONDITIONS: ANCA Associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Intervention Model Description: Subjects with normalized CD5+ B cells are thought to be at lower risk and relapse, and therefore may not need maintenance immunosuppression. The subjects in that group will be randomized to either maintenance immunosuppression vs close clinical observation without maintenance immunosuppression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- low CD5+ /on maintenance (Active Comparator): Subjects in remission with Cluster of Differentiation 19 positive (CD19+) CD5+ lower than 43% will continue on maintenance immunosuppression (Maintenance Therapy Group)- no randomization.
  Interventions: Device: ENUMERATION OF CD5+ B Cells
- high CD5/ on maintenance (Active Comparator): Subjects in remission with CD19+CD5+ 43% or greater, randomized to continue on maintenance immunosuppression (Maintenance Therapy Group)
  Interventions: Device: ENUMERATION OF CD5+ B Cells
- high CD5 / NO maintenance (Experimental): Subjects in remission with CD19+CD5+ 43% or greater , randomized to NO maintenance immunosuppression (NO Maintenance Therapy Group)
  Interventions: Device: ENUMERATION OF CD5+ B Cells

INTERVENTIONS:
Device: ENUMERATION OF CD5+ B Cells — A blood test is done to assess what percentage of CD5+ is present within CD19+. The result is then used to guide choice of arm.

SUMMARY:
ANCA vasculitis is a pauci-immune systemic small vessel vasculitis. The anti-neutrophilic cytoplasmic antibodies (ANCA) are pathogenic and cause disease by activating neutrophils which damage blood vessels. CD means "cluster of differentiation" . CD5 is a type I transmembrane protein found on T cells, thymocytes, and some B cells. Cluster of Differentiation 20 (CD20) is a type III transmembrane protein found on B cells. The investigators previously detected an association between recovery of Interleukin 10 (IL-10)-secreting CD20+ and CD5+ regulatory B cells after immunotherapy (with rituximab and corticosteroids) and decreased risk of subsequent relapse in patients with ANCA-vasculitis. The investigators hypothesize that patients with complete reconstitution of a functional regulatory B cell repertoire after induction therapy are at low risk of relapse and may be monitored conservatively without further immunotherapy. The investigators will test this hypothesis through a proof of concept randomized controlled study. Patients with normalization of CD5+ regulatory B cells will be randomized to maintenance therapy with rituximab vs. close observation without immunosuppression. Patients whose peripheral CD5+ regulatory B cells remain low after induction therapy (who are at higher risk of relapse), will receive maintenance immunosuppression with rituximab. Patients needing or randomized to maintenance therapy who are unable to receive rituximab will receive azathioprine or mycophenolate mofetil, two standard alternative medications for maintenance immunosuppression.

DETAILED DESCRIPTION:
The goal of this study is to test the hypothesis that, in ANCA vasculitis, use of CD5+ B cells at the time of B cell reconstitution in the peripheral blood can be used to stratify patients between those with low % CD5+ B cells at greater risk of relapse who would need maintenance immunosuppression and those with normalized CD5+ B cells who would be at lower risk of relapse, and therefore may not need maintenance immunosuppression. The latter group will be randomized to either maintenance immunosuppression vs close clinical observation without maintenance immunosuppression. This study is not designed to evaluate the efficacy of new therapies in ANCA vasculitis. The treatment regimen used in the proposed study are routinely used in the treatment of patients with ANCA vasculitis and considered standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-85 years old.
* ANCA Glomerulonephritis (GN) or vasculitis per Chapel Hill Consensus Criteria, with documented current or previously positive Myeloperoxidase (MPO)- or Proteinase 3 (PR3)-ANCA by ELISA test. Patients with biopsy-proven, pauci-immune crescentic glomerulonephritis are eligible if they have a positive ANCA test by immunofluorescent microscopy (IIFM).
* Patients must be in complete remission for at least 1 month and after AT LEAST 3 MONTHS of induction of therapy with corticosteroids and rituximab (either 1000 mg IV x 2 or 375 mg/m2 IV x 4) OR corticosteroids and cyclophosphamide (monthly IV or daily oral doses). They must be on no more than 5 mg daily of oral prednisone or equivalent. Complete remission is defined as a Birmingham Vasculitis Activity Score (BVAS) score = 0.
* Patients may be ANCA negative or positive at randomization.
* B cells are not depleted anymore: B cell recovery reaches 1% CD19+ B cells (enough to allow determination of CD5+ B cells with confidence).

Exclusion Criteria:

* Patients who have had ≥ 2 relapses (defined as recurrence of any signs or symptoms attributable to active vasculitis) previously as patients with multiple prior relapses may be at higher risk of future relapse and require maintenance therapy
* Patients with persistent low-grade disease activity ("grumbling" disease defined as BVAS > 0 and ≤ 3)
* Patients with active systemic infections or deep space infections within the 3 months prior to screening.
* Patients participating in another clinical trial mandating maintenance therapy
* Patients with drug-induced ANCA vasculitis (e.g. levamisole-adulterated cocaine)
* Active tuberculosis, human immunodeficiency virus (HIV), hepatitis C virus or hepatitis B virus infections
* For women of child-bearing potential, pregnancy, breastfeeding, unwillingness or inability to comply with effective contraception
* Inability to come to scheduled visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vimal Derebail, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and data use/sharing agreement with UNC.

REFERENCES:
- [Result] Guillevin L, Pagnoux C, Karras A, Khouatra C, Aumaitre O, Cohen P, Maurier F, Decaux O, Ninet J, Gobert P, Quemeneur T, Blanchard-Delaunay C, Godmer P, Puechal X, Carron PL, Hatron PY, Limal N, Hamidou M, Ducret M, Daugas E, Papo T, Bonnotte B, Mahr A, Ravaud P, Mouthon L; French Vasculitis Study Group. Rituximab versus azathioprine for maintenance in ANCA-associated vasculitis. N Engl J Med. 2014 Nov 6;371(19):1771-80. doi: 10.1056/NEJMoa1404231. PMID 25372085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Individuals who signed informed consent and then completed all baseline measurement procedures and remained eligible were considered enrolled and were randomized. One consented participant experienced a Serious Adverse Event and was withdrawn before randomization and another consented participant was screen failed because they were not in remission.
Groups:
- Low CD5+ /on Maintenance: Participants in remission with Cluster of Differentiation (CD)19+CD5+ lower than 43% will continue on maintenance immunosuppression (Maintenance Therapy Group)- no randomization.
  ENUMERATION OF CD5+ B Cells: A blood test is done to assess what percentage of CD5+ is present within CD19+. The result is then used to guide choice of arm.
- High CD5/ on Maintenance: Participants in remission with Cluster of Differentiation 19 positive (CD19+)CD5+ 43% or greater, randomized to continue on maintenance immunosuppression (Maintenance Therapy Group)
  ENUMERATION OF CD5+ B Cells: A blood test is done to assess what percentage of CD5+ is present within CD19+. The result is then used to guide choice of arm.
- High CD5 / NO Maintenance: Participants in remission with CD19+CD5+ 43% or greater , randomized to NO maintenance immunosuppression (NO Maintenance Therapy Group)
  ENUMERATION OF CD5+ B Cells: A blood test is done to assess what percentage of CD5+ is present within CD19+. The result is then used to guide choice of arm.
Period: Overall Study
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance
Started | 1 | 4 | 2
Completed | 1 | 2 | 2
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- High CD5/ on Maintenance: Participants in remission with CD19+CD5+ 43% or greater, randomized to continue on maintenance immunosuppression (Maintenance Therapy Group)
  ENUMERATION OF CD5+ B Cells: A blood test is done to assess what percentage of CD5+ is present within CD19+. The result is then used to guide choice of arm.
- Total: Total of all reporting groups
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance | Total
Number analyzed (Participants) | 1 | 4 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4
  >=65 years | 0 | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 0 | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 0 | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 1 | 4 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 4 | 2 | 7
Anti-Neutrophilic Cytoplasmic Antibodies (ANCA) Positive at Enrollment [Count of Participants; unit: Participants] | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse
Description: The primary outcome measure is time to first relapse defined as recurrence of any signs or symptoms attributable to active vasculitis after a period of complete remission, with at least 2 minor or 1 major item on the BVAS score (BVAS≥2). Per protocol, complete remission is defined as a BVAS score = 0. Birmingham Vasculitis Activity Score (BVAS, range 0-64). The total score is composed of 34 predefined items, units on a scale, grouped into 9 organ systems. Each item carries a weight from 1-3, depending on disease severity. A score of 0 indicates no disease activity; a higher score indicates worsening disease.
Time Frame: from complete remission to end of study, approximately 2 years
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance
Number analyzed (Participants) | 1 | 4 | 2
months | 7.1 (0) | NA (NA) — No participants in this Arm/Group experienced relapse | NA (NA) — No participants in this Arm/Group experienced relapse

2. Secondary Outcome: Number of Participants Who Experience Relapse
Description: Relapse in each group was determined using the Birmingham Vasculitis Activity Score for Wegener's Granulomatosis(BVAS, range 0-64). The total score is composed of 34 predefined items grouped into 9 organ systems. Each item has a specified weight of either 3 or 1, depending on whether it reflects major or minor disease activity. A score of 0 indicates no disease activity; a higher score indicates worsening disease. Per protocol relapse is defined as BVAS >/= 2; however for reporting purposes relapse was defined as BVAS >/= 1 because the participant was treated based on the clinical relapse.
Time Frame: from complete remission to end of study, approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance
Number analyzed (Participants) | 1 | 4 | 2
Participants | 1 | 0 | 0

3. Secondary Outcome: Frequency of Relapse
Description: Frequency, as determined by number of relapse in each group. Per protocol relapse is defined as BVAS >/= 2; however for reporting purposes relapse was defined as BVAS >/= 1 because the participant was treated based on the clinical relapse.
Time Frame: from complete remission to end of study, approximately 2 years
Measure: Number; unit: relapse
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance
Number analyzed (Participants) | 1 | 4 | 2
relapse | 1 | 0 | 0

4. Secondary Outcome: Severity of Relapse
Description: Severity of relapse as determined by number of major relapse in each group. Major relapse is defined as involving a major organ
Time Frame: from complete remission to end of study, approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance
Number analyzed (Participants) | 1 | 4 | 2
Participants
  Major | 0 | 0 | 0
  Minor | 1 | 0 | 0
  No relapse | 0 | 4 | 2

5. Secondary Outcome: Time to Positive ANCA
Description: For participants who had a negative ANCA test, time to positive ANCA
Time Frame: from first negative ANCA test since start of study , if applicable- to end of study, maximum two years, as applicable
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance
Number analyzed (Participants) | 1 | 4 | 2
months | NA (NA) — ANCA test did not become positive. | NA (NA) — No data are reported because two were ANCA-positive at enrollment and two never became positive. | NA (NA) — ANCA test did not become positive.

6. Secondary Outcome: Frequency of Infections
Description: Frequency as determined by the number of infections
Time Frame: from remission to end of study, approximately 2 years
Measure: Number; unit: infections
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance
Number analyzed (Participants) | 1 | 4 | 2
infections | 0 | 0 | 1

7. Secondary Outcome: Number of Infections, Categorized by Severity
Description: number of mild/moderate/severe infections
Time Frame: from remission to end of study, approximately 2 years
Measure: Number; unit: infection
Groups:
- Non-Randomized: Participants who signed informed consent but could not be randomized.
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance | Non-Randomized
Number analyzed (Participants) | 1 | 4 | 2 | 2
infection
  Mild | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0

8. Secondary Outcome: Time to Interleukin (IL)-10 Secreting B Regulatory Cells > 45% or CD5+ B Cells > 43% of Total B Cells
Description: Time to IL-10 secreting B regulatory cells > 45% or CD5+ B cells > 43% of total B cells
Time Frame: from enrollment to end of study, approximately 2.5 to 3 years
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance
Number analyzed (Participants) | 1 | 4 | 2
months | NA (NA) — The participant who experienced relapse did not have IL-10 secreting B regulatory cells > 45% or CD5+ B cells > 43% of total B cells. | NA (NA) — No participants experienced relapse. | NA (NA) — No participants experienced relapse.

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, up to 2 years
Arm/Group | Low CD5+ /on Maintenance | High CD5/ on Maintenance | High CD5 / NO Maintenance | Non-Randomized
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/4 | 2/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low CD5+ /on Maintenance (N=1) | High CD5/ on Maintenance (N=4) | High CD5 / NO Maintenance (N=2) | Non-Randomized (N=2)
Intracranial mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low CD5+ /on Maintenance (N=1) | High CD5/ on Maintenance (N=4) | High CD5 / NO Maintenance (N=2) | Non-Randomized (N=2)
Prolonged fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Post Rituxan infusion
Pruritic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reaction to Shingrix vaccination (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncopal episode resulting in fall with head trauma (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right knee swollen and hot to touch (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Similar to gout flare symptoms
Increase in right hydrocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilateral leg weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Belching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture of left radius (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal urinalysis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon nodules (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
"Trigger finger" (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain at vaccination site (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small left eye hemorrhage at inner area (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart burn when lying down (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma skin lesion on right arm above elbow-removed (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Further removal of squamous cell carcinoma on right arm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right foot Planter's wart removal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff tear left shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subsequent to shingles vaccine
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain from frozen shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low vitamin B (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
rituximab infusion reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03906227/Prot_SAP_001.pdf
  • Informed Consent Form (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT03906227/ICF_000.pdf